CLINICAL TRIAL: NCT00219323
Title: Long-Term Study of IGE025 in Moderate to Severe Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025A1307
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: Asthma, IgE, Omalizumab
MeSH Terms: conditions — Asthma; Epilepsy, Idiopathic Generalized | interventions — Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
This study will evaluate the safety and efficacy of omalizumab up to 48 weeks in adult patients with moderate to severe bronchial asthma.

THIS STUDY IS NOT ENROLLING PATIENTS IN THE UNITED STATES

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthma patients
* Inadequately controlled patients

Exclusion Criteria:

* - History of severe anaphylactoid or anaphylactic reactions
* Previous treatment with omalizumab
* History of cancer or cancer

Other protocol-defined exclusion criteria may apply.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2003-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Safety of omalizumab

SECONDARY OUTCOMES:
Pulmonary function parameters measured by spirometer
Morning and evening peak expiratory flow (PEF)
Symptoms score, treatment score, activities of daily living score, nighttime sleep score, and asthma score

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals Japan
Locations (1):
- This study is not being conducted in the United States, Tokyo, Japan